Title: Effect of Sport Education in University Required PE on Students'
Perceived Physical Literacy and Physical Activity Level

NCT number: NCT03888885

Date: 12/9/2021



### The Chinese University of Hong Kong

#### **Consent Form**

Project title: Effects of Sport Education Intervention in University Required Physical

**Education: Cluster Randomized Trial of Students' Perceived Physical** 

**Literacy and Physical Activity Levels** 

Investigator: Choi Siu Ming

Department of Sports Science & Physical Education (SSPE)

Supervisor: Sum Kim Wai, Raymond

Department of Sports Science & Physical Education (SSPE)

First of all, thank you for your interest to take part in this project. Please take your time to review this consent form and discuss any questions you may have, or words you do not clearly understand, with the investigator or staff.

# **Purpose of the Study**

The purpose of this study is to examine the effectiveness of Sport Education model delivered in the required physical education lessons at the university level on students perceived physical literacy and physical activity levels.

#### **Study Procedures**

Upon receiving your consent, you will be requested to complete a set of questionnaires consisting Empowering and Disempowering Motivational Climate Questionnaire in Physical Education (Milton et al., 2018), The Situational Motivation Scale (Guay et al., 2000), Perceived Physical Literacy Instrument (Sum et al., 2016), The Physical Activity Enjoyment Scale (Motl et al., 2001), International Physical Activity Questionnaire – short form (Booth et al., 2000). Some demographic information such as age, gender, height, weight, studying faculty and sports participating levels will also be collected. It takes about 15 minutes to complete. A sub-sample of 128 participants (8 students in each class) will be randomly selected to wear accelerometers to measure their objective physical activity levels for at least 8 hours per day, in 7 consecutive days at the same period of time. During the intervention period, all lessons will be videotaped and coded by System for Observing Fitness Instruction Time (McKenzie, Sallis, & Nader, 1992). You will be requested to complete the questionnaire and the sub-sample group needs to wear the accelerometer for one week at the end of intervention and at the 3rd week post intervention.

#### **Confidentiality**

Your participation in this study will be strictly confidential. Your real name will not be used in this study. No identifying information and name will be used and revealed in any written reports or publications. All findings in this study will be reported in aggregate form with no identifying information. All data will be kept by the researcher for 12 months beyond the end of the study.

## **Voluntary Participation**

Your participation is completely voluntary, and you may withdraw your participation at any time during the process, either temporarily or permanently.

Should any questions arise at any point during the study, please do not hesitate to contact me at +852 3943 6079 (office) or my supervisor at +852 3943 6091 (office).

## **Statement of Consent - Informed Consent Form for Adults**

I have read the above information and have received answers to any questions I asked. I understood the nature of this study and agree that the information collected will be kept by the researcher for 12 months beyond the end of the study.

| By signing below, I indi | cate my consent to: | | |
|---|---|---|---|
| ☐ Take part in the study | <b>7.</b> | | |
| ☐ Agree to the video-re | cording / audio-recording duri | ng the procedure. | |
| Signature of Participant: | | D | ate: |
| | (Printed Name: | ) | |
| Signature of Person Obtaining Consent: | | D | ate: |
| | (Printed Name: | ) | |